CLINICAL TRIAL: NCT06154512
Title: A Real-world, Multi-center, Prospective, Observational Study for Paroxysmal Nocturnal Haemoglobinuria (PNH) in China
Brief Title: A Real-world, Multi-center, Prospective, Observational Study for PNH in China
Acronym: ReWoPNH
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D7414R00001
Record Dates: First submitted 2023-10-30; First posted 2023-12-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — only collect data from patients' medical history, do not collect patient biospecimen directly.

SUMMARY:
As a rare disease listed in the First Catalogue of Rare Diseases in China (National Health Commission of the People's Republic of China, 2019), PNH is poorly studied in China subse-quently leading to the inadequate elucidation of disease characteristics and clinical outcomes. Eculizumab was recently approved by NMPA. The availability of Eculizumab in China pro-vides people living with PNH with a new treatment option that can reduce disease symptoms and prevent the dysregulated complement system from causing further damage. A Phase Ⅳ study is necessary to understand the natural history of disease and the clinical outcomes with different medical interventions.

DETAILED DESCRIPTION:
Paroxysmal nocturnal hemoglobinuria (PNH) is an ultra-rare and life-threatening acquired disorder of the pluripotent hematopoietic stem cell and therefore can affect erythrocytes, leukocytes, thrombocytes and probably some endothelial cells. These hematopoietic stem cells have acquired a somatic mutation in the phosphatidylinositol glycan class A (PIG-A) This gene is required for the synthesis of the glycosyl phosphatidyl-inositol (GPI) anchor, which is necessary to attach some proteins to the blood cell membrane. Therefore, a lack of two important complement regulatory proteins is observed on the cell surface: 'decay-accelerating factor' (DAF), also called 'CD55' and 'membrane inhibitor of reactive lysis' (MIRL), also called 'CD59' Thus, red blood cells are more vulnerable to the attack by the complement activation product MAC (complement membrane attack complex). This leads to a complement-mediated intravascular hemolysis. The predisposition of venous thrombosis, hemolytic anemia, complete thrombocytopenia, and thrombosis are the three main characteristics of the disease. Its incidence is not really known but estimated at 0.1~0.6/100 000 per-sons/yr, and prevalence is estimated at 1~4 cases/100,000 persons/yr. PNH was listed in the First Catalogue of Rare Diseases in China, and its incidence was previously reported to be 1/100,000 persons/year, peak onset age 20~40 years.

PNH can be classified into 3 different forms: classical PNH, PNH associated with aplastic anemia (PNH-AA), and subclinical PNH, based on clinical features, bone marrow characteristics, and the size of the mutant clone. The traditional treatment of PNH is still aimed at "protecting" the PNH clone, reducing complement attack and destruction, and alleviating hemolysis with symptomatic supportive therapy. In acute hemolytic episodes, could be administered adrenal glucocorticoids, complemented by cell membrane stabilizers, folic acid, and alkaline drugs. In case of PNH-AA syndrome, treatment with androgens and immunosuppressants may be used; anticoagulation and heparin therapy should be given for the occurrence of thrombosis; other symptomatic supportive treatments include transfusion of red blood cells and platelets if necessary as well as antibacterial drugs in case of infection. Bone marrow transplantation is the only curative therapy for PNH presupposes, but patient need to achieve complete remission with chemotherapy first and a suitable donor is needed.

Besides supportive care, global guidance/consensus also recommend C5 complement inhibitor Eculizumab as a treatment method, and its use could significantly improve 5-year survival rate to 95.5%. Eculizumabis a humanized, first-in-class, anti-C5 antibody that binds with high affinity to C5 and blocks the terminal complement-C5a and C5b-9 formation, reducing the chronic uncontrolled complement activation and its consequences. Eculizumab has been approved for PNH by National Medical Products Administration in August, 2022.

ELIGIBILITY:
Inclusion Criteria

1. Patients of any age;
2. Diagnosed PNH with detected proportion of PNH clone cells of at least 1%;
3. Patient or patient's family must be willing and able to give written informed consent.

Exclusion Criteria

1. Current or previous treatment with a non-eculizumab complement inhibitor;
2. Patients in other PNH clinical trials.
3. Unable to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study Population:
  Number of patients (estimate): 1000; Inclusion Criteria
  1. Patients of any age;
  2. Diagnosed PNH with detected proportion of PNH clone cells of at least 1%;
  3. Patient or patient's family must be willing and able to give written informed consent.
  Exclusion Criteria
  1. Current or previous treatment with a non-eculizumab complement inhibitor;
  2. Patients in other PNH clinical trials.
  3. Unable to give written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 724 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Hemolysis：Concentration of LDH changes at each visit from base-line, of all patients | 12 months
  To characterize the progression of PNH
Number and percentage of patients with thrombosis within follow-up | 12 months
  To characterize the progression of PNH
average number of units of packed RBCs transfused per month, of all patients | 12 months
  To characterize the progression of PNH
Number and percentage of patients with renal failure within follow-up | 12 months
  To characterize the progression of PNH
Number and percentage of patients with pulmonary hypertension within follow-up | 12 months
  To characterize the progression of PNH

SECONDARY OUTCOMES:
Number and percentage of patients with each symptom of interest within follow-up | 12 months
  To describe clinical characteristics of patients with PNH in China
Demographics at baseline of all patients | baseline
  To describe clinical characteristics of patients with PNH in China
Number and percentage of patients receiving each type of treatment method at baseline and each visit within follow up, including glucocorticoid, red blood cell transfusion, other supportive treatment, bone marrow transplant, eculizumab, of all patients | 12 months
  To describe the treatment pattern of PNH in China
All serious adverse events (SAEs)of PNH among eculizumab-treated patients | 12 months
  To describe the safety of Eculizumab treatment via Serious Adverse Events
Standard descriptive statistics of pregnancy status | 12 months
  To describe clinical characteristics of patients with PNH in China
Standard descriptive statistics of lactation status | 12 months
  To describe clinical characteristics of patients with PNH in China
Standard descriptive statistics of PNH classification | 12 months
  To describe clinical characteristics of patients with PNH in China
Standard descriptive statistics of flow cytometry results | 12 months
  To describe clinical characteristics of patients with PNH in China

OTHER OUTCOMES:
Concentration of LDH changes at each visit from base-line of PNH among eculizumab-treated patients | 12 months
  Exploratory objective: To characterize the progression of PNH among eculizumab-treated patients
Number and percentage of patients with thrombosis within follow up among eculizumab-treated patients | 12 months
  Exploratory objective: To characterize the progression of PNH among eculizumab-treated patients
average number of units of packed RBCs transfused per month within 12 months v | 12 months
  Exploratory objective: To characterize the progression of PNH among eculizumab-treated patients
Number and percentage of patients with renal failure within follow up among eculizumab-treated patients | 12 months
  Exploratory objective: To characterize the progression of PNH among eculizumab-treated patients
Number and percentage of patients with pulmonary hypertension (PH) within follow up among eculizumab-treated patients | 12 months
  Exploratory objective: To characterize the progression of PNH among eculizumab-treated patients

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - Research Site, Hefei, Anhui
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Nanning, Guangxi
  - Research Site, Guiyang, Guizhou
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Harbin, Heilongjiang
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Nantong, Jiangsu
  - Research Site, Xuzhou, Jiangsu
  - Research Site, Nanchang, Jiangxi
  - Research Site, Changchun, Jilin
  - Research Site, Shenyang, Liaoning
  - Research Site, Jinan, Shandong
  - Research Site, Qingdao, Shandong
  - Research Site, Zibo, Shandong
  - Research Site, Linyi, Shangdong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Kunming, Yunnan
  - Research Site, Hangzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/